CLINICAL TRIAL: NCT02321228
Title: Early Salpingectomy (Tubectomy) With Delayed Oophorectomy to Improve Quality of Life as Alternative for Risk Reducing Salpingo-oophorectomy in BRCA1/2 Gene Mutation Carriers
Brief Title: Early Salpingectomy (Tubectomy) With Delayed Oophorectomy in BRCA1/2 Gene Mutation Carriers
Acronym: TUBA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Nijmegen (Other)
Responsible Party: Principal Investigator, Joanne A. de Hullu, MD, PhD, MD, PhD, gynecologic oncologist, principal clinician, University Medical Center Nijmegen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL50048.091.14
Record Dates: First submitted 2014-12-11; First posted 2014-12-22 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: BRCA1 Gene Mutation; BRCA2 Gene Mutation; Ovarian Cancer
Keywords: Salpingectomy; Delayed oophorectomy; Salpingo-oophorectomy; Quality of life; Ovarian cancer; BRCA
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Salpingectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Salpingectomy with delayed oophorectomy (Experimental): Female BRCA mutation carriers can opt for early salpingectomy upon completion of childbearing, followed by second stage oophorectomy delayed for five years beyond current guideline ages for risk-reducing salpingo-oophorectomy (i.e. age 40-45 for BRCA1 mutation carriers and 45-50 for BRCA mutation carriers).
  Interventions: Procedure: Salpingectomy with delayed oophorectomy
- Risk-reducing salpingo-oophorectomy (Active Comparator): Female BRCA mutation carriers can opt for standard risk-reducing salpingo-oophorectomy at current guideline ages (age 35-40 for BRCA1 mutation carriers and age 40-45 for BRCA2 mutation carriers).
  Interventions: Procedure: Risk-reducing salpingo-oophorectomy

INTERVENTIONS:
Procedure: Salpingectomy with delayed oophorectomy — Early salpingectomy upon completions of childbearing with postponement of oophorectomy until between 40 and 45 in BRCA1 mutation carriers and between age 45 and 50 in BRCA2 mutation carriers.
  Other Names: Tubectomy with delayed oophorectomy
  Arms: Salpingectomy with delayed oophorectomy
Procedure: Risk-reducing salpingo-oophorectomy — This is the current guideline procedure, usually performed between age 35 and 40 in BRCA1 mutation carriers and between age 40 and 45 in BRCA2 mutation carriers.
  Other Names: Bilateral prophylactic salpingo-oophorectomy
  Arms: Risk-reducing salpingo-oophorectomy

SUMMARY:
The purpose of this study is to determine whether an innovative preventive strategy, consisting of early salpingectomy upon completion of childbearing with delayed oophorectomy beyond current guideline age, improves menopause-related quality of life without significantly increasing ovarian cancer incidence in comparison to current standard salpingo-oophorectomy in female BRCA1/2 mutation carriers.

DETAILED DESCRIPTION:
Eligible women will choose for the innovative or standard risk-reducing option themselves.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women with a documented BRCA1 and/or BRCA2 germline mutation
* Age 25-40 years for BRCA1 mutation carriers, 25-45 years for BRCA2
* Childbearing completed
* Presence of at least one fallopian tube
* Participants may have a personal history of non-ovarian malignancy

Exclusion Criteria:

* Postmenopausal status (natural menopause or due to (cancer) treatment)
* Wish for second stage oophorectomy within two years after salpingectomy (if clear at enrollment)
* Legally incapable
* Prior bilateral salpingectomy
* A personal history of ovarian, fallopian tube or peritoneal cancer
* Evidence of malignant disease at enrollment
* Treatment for malignant disease at enrollment
* Inability to read or speak Dutch

BRCA mutation carriers who opt for salpingectomy but who do not want to postpone the oophorectomy beyond the guideline age will undergo similar follow-up but do not contribute to the 510 inclusions we need

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 510 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Menopause-related quality of life | Up to 5 years after last surgery
  Measured by the Greene Climacteric Scale

SECONDARY OUTCOMES:
General quality of life | Up to 15 years after last surgery
  measured by several questionnaires
Quality of life related items | Up to 15 years after last surgery
  i.e. sexual functioning, cancer worry, satisfaction with decision
Surgery-related complications | 6 weeks after each surgery
  Surgery-related complications
Histopathologic findings of removed fallopian tubes and ovaries | 6 weeks after each surgery
  - Histopathologic findings of removed fallopian tubes and ovaries
Cardiovascular risk factors | Up to 5 years after last surgery
  Limited physical examination: blood pressure, BMI, waist-hip ratio Blood sample Questionnaires on cardiovascular risk factors and diseases
Incidence of cardiovascular diseases | Up to 15 years after last surgery
  i.e. waist-hip circumference, Fasting blood sample
Incidence of ovarian cancer | Up to 15 years after last surgery
  Incidence of ovarian cancer (cancer of tubes, ovaries and/or peritoneal cancer)
Incidence of breast cancer | Up to 15 years after last surgery
  Incidence of breast cancer
Cost-effectiveness of innovative preventive strategy | 10 years after last surgery
  Costs per quality adjusted life year (QALY)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne A de Hullu, MD, PhD, Principal Investigator — University Medical Center Nijmegen; Rosella PM Hermens, PhD, Principal Investigator — Scientific Institute for Quality of Healtcare, UMCNijmegen; Nicoline Hoogerbrugge, MD, PhD, Principal Investigator — University Medical Center Nijmegen
Locations (13):
- Netherlands (13):
  - Maastricht University Medical Center, Maastricht, Limburg
  - Catharina Hospital, Eindhoven, North Brabant
  - Elisabeth-TweeSteden Hospital, Tilburg, North Brabant
  - Netherlands Cancer Institute / Antoni van Leeuwenhoek Hospital, Amsterdam, North Holland
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - Academic Medical Center, Amsterdam
  - VU University Medical center, Amsterdam
  - University Medical Center Groningen, Groningen
  - Medical Center, Leeuwarden
  - Radboudumc, Nijmegen
  - University Medical Center Utrecht, Utrecht
  - Maxima Medical Center, Veldhoven

REFERENCES:
- [Derived] van Bommel MHD, Steenbeek MP, IntHout J, Hermens RPMG, Hoogerbrugge N, Harmsen MG, van Doorn HC, Mourits MJE, van Beurden M, Zweemer RP, Gaarenstroom KN, Slangen BFM, Brood-van Zanten MMA, Vos MC, Piek JM, van Lonkhuijzen LRCW, Apperloo MJA, Coppus SFPJ, Prins JB, Custers JAE, de Hullu JA. Cancer worry among BRCA1/2 pathogenic variant carriers choosing surgery to prevent tubal/ovarian cancer: course over time and associated factors. Support Care Cancer. 2022 Apr;30(4):3409-3418. doi: 10.1007/s00520-021-06726-4. Epub 2022 Jan 8. PMID 34997316
- [Derived] Steenbeek MP, Harmsen MG, Hoogerbrugge N, de Jong MA, Maas AHEM, Prins JB, Bulten J, Teerenstra S, van Bommel MHD, van Doorn HC, Mourits MJE, van Beurden M, Zweemer RP, Gaarenstroom KN, Slangen BFM, Brood-van Zanten MMA, Vos MC, Piek JMJ, van Lonkhuijzen LRCW, Apperloo MJA, Coppus SFPJ, Massuger LFAG, IntHout J, Hermens RPMG, de Hullu JA. Association of Salpingectomy With Delayed Oophorectomy Versus Salpingo-oophorectomy With Quality of Life in BRCA1/2 Pathogenic Variant Carriers: A Nonrandomized Controlled Trial. JAMA Oncol. 2021 Aug 1;7(8):1203-1212. doi: 10.1001/jamaoncol.2021.1590. PMID 34081085
- [Derived] Harmsen MG, Arts-de Jong M, Hoogerbrugge N, Maas AH, Prins JB, Bulten J, Teerenstra S, Adang EM, Piek JM, van Doorn HC, van Beurden M, Mourits MJ, Zweemer RP, Gaarenstroom KN, Slangen BF, Vos MC, van Lonkhuijzen LR, Massuger LF, Hermens RP, de Hullu JA. Early salpingectomy (TUbectomy) with delayed oophorectomy to improve quality of life as alternative for risk-reducing salpingo-oophorectomy in BRCA1/2 mutation carriers (TUBA study): a prospective non-randomised multicentre study. BMC Cancer. 2015 Aug 19;15:593. doi: 10.1186/s12885-015-1597-y. PMID 26286255